CLINICAL TRIAL: NCT03879135
Title: A Phase 3b, Prospective, Open-Label, Uncontrolled, Multicenter Study on Long-Term Safety and Efficacy of rVWF in Pediatric and Adult Subjects With Severe Von Willebrand Disease (VWD)
Brief Title: A Study of Recombinant Von Willebrand Factor (rVWF) in Pediatric and Adult Participants With Severe Von Willebrand Disease (VWD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SHP677-304; 2018-003453-16 (EudraCT Number)
Record Dates: First submitted 2018-12-20; First posted 2019-03-18 (Actual); Results first posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Von Willebrand Disease (VWD)
MeSH Terms: conditions — von Willebrand Diseases | interventions — Factor VIII; F8 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- On-Demand (Experimental): Participants will receive recombinant von Willebrand factor (rVWF) (with or without ADVATE).
  Interventions: Biological: rVWF; Biological: rFVIII
- Prophylaxis (Experimental): Participants will receive recombinant von Willebrand factor (rVWF).
  Interventions: Biological: rVWF; Biological: rFVIII

INTERVENTIONS:
Biological: rVWF — Recombinant von Willebrand factor
  Other Names: Vonvendi; Vonicog alfa
Biological: rFVIII — Recombinant Factor VIII
  Other Names: Octocog alfa; ADVATE

SUMMARY:
The main aim of the study is to check effectiveness of rVWF (vonicog alfa) prophylaxis based on the annualized bleeding rate (ABR) of spontaneous (not related to trauma) bleeding episodes in pediatric and adult participants during the first 12 months on study treatment.

The participants will be treated with rVWF for a maximum of 3 years. Their von Willebrand Disease will be treated according to Investigational product (IP) dosing directions.

ELIGIBILITY:
Inclusion Criteria:

The participant will not be considered eligible for the study without meeting all of the criteria below.

Participants who have completed Study 071301 or Study 071102 (or participants who have completed the surgery arm treatment in Study 071102 and want to continue to receive on-demand (OD) treatment) and are willing to immediately transition into this study, must meet the following 2 criteria to be eligible for this study:

* If female of childbearing potential, has a negative blood/urine pregnancy test at screening and agrees to employ highly effective birth control measures for the duration of the study.
* Participant and/or legally authorized representative is willing and able to comply with the requirements of the protocol.

New participants (Cohort 4) who meet the above 2 and ALL the following additional criteria are eligible for this study:

- Participant has a documented diagnosis of severe von Willebrand disease (VWD) (baseline von Willebrand factor: Ristocetin cofactor (VWF:RCo) <20 International Units per deciliter [IU/dL]) with a history of requiring substitution therapy with von Willebrand factor (vWF) concentrate to control bleeding:

* Type 1 (VWF:RCo <20 IU/dL) or,
* Type 2A (as verified by multimer pattern), Type 2B (as diagnosed by genotype), Type 2M or,
* Type 3 (Von Willebrand factor antigen (VWF:Ag) less than or equal to (<=) 3 IU/dL).

Diagnosis is confirmed by genetic testing and multimer analysis, documented in participant history or at screening.

* Participant has been receiving OD therapy with VWF products for at least 12 months, and prophylactic treatment is recommended by the investigator.
* Participant has greater than or equal to (>=) 3 documented spontaneous bleeds (not including menorrhagia) requiring VWF treatment during the past 12 months.
* Participant has available records that reliably evaluate type, frequency, and treatment of bleeding episodes for at least 12 months preceding enrollment; up to 24 months of retrospective data should be collected if available.
* Participant is >=12 years old at the time of screening and has a body mass index >=15 but <40 kilogram per meter square (kg/m^2).

Exclusion Criteria:

The participant will be excluded from the study if any of the following exclusion criteria are met.

* The participant has been diagnosed with Type 2N VWD, pseudo VWD, or another hereditary or acquired coagulation disorder other than VWD (eg, qualitative and quantitative platelet disorders or elevated prothrombin time (PT)/international normalized ratio [INR] >1.4).
* The participant has a history or presence of a VWF inhibitor at screening.
* The participant has a history or presence of a Factor VIII (FVIII) inhibitor with a titer >=0.4 Bethesda units (BU) (by Nijmegen modified Bethesda assay) or >=0.6 BU (by Bethesda assay).
* The participant has a known hypersensitivity to any of the components of the study drugs, such as mouse or hamster proteins.
* The participant has a medical history of immunological disorders, excluding seasonal allergic rhinitis/conjunctivitis, mild asthma, food allergies, or animal allergies.
* The participant has a medical history of a thromboembolic event.
* The participant is human immunodeficiency virus (HIV) positive with an absolute Helper T cell (CD4) count <200/cubic millimeters (mm^3).
* The participant has been diagnosed with significant liver disease per investigator's medical assessment of the participant's current condition or medical history or as evidenced by, but not limited to any of the following: serum alanine aminotransferase (ALT) greater than 5 times the upper limit of normal; hypoalbuminemia; portal vein hypertension (eg, presence of otherwise unexplained splenomegaly, history of esophageal varices) or liver cirrhosis classified as Child-Pugh class B or C.
* The participant has been diagnosed with renal disease, with a serum creatinine (CR) level >=2.5 milligrams per deciliter (mg/dL).
* The participant has a platelet count <100,000/milliliter (mL) at screening.
* The participant has been treated with an immunomodulatory drug, excluding topical treatment (eg, ointments, nasal sprays), within 30 days prior to signing the informed consent (or assent, if appropriate).
* The participant is pregnant or lactating at the time of enrollment.
* The participant has cervical or uterine conditions causing menorrhagia or metrorrhagia (including infection, dysplasia).
* The participant has participated in another clinical study involving another investigational product (IP) or investigational device within 30 days prior to enrollment or is scheduled to participate in another clinical study involving an IP or investigational device during the course of this study.
* The participant has a progressive fatal disease and/or life expectancy of less than 15 months.
* For new OD participants, the participant is scheduled for a surgical intervention.
* The participant is identified by the investigator as being unable or unwilling to cooperate with study procedures.
* The participant has a mental condition rendering him/her unable to understand the nature, scope and possible consequences of the study and/or evidence of an uncooperative attitude.
* The participant is member of the study team or in a dependent relationship with one of the study team members which includes close relatives (i.e., children, partner/spouse, siblings and parents) as well as employees.

Delay criteria Only for Cohort 4, if the participant presents with an acute bleeding episodes or acute illness (eg, influenza, flu-like syndrome, allergic rhinitis/conjunctivitis, and non-seasonal asthma) the screening visit will be postponed until the participant has recovered. For all other participants, end of study (EOS) visit for 071102 or 071301 will be completed per protocol and the completed EOS in Study 071102 or 071301 will also serve as the screening visit for this continuation study (SHP677-304).

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (31):
- United States (8):
  - Arkansas Children's Hospital Research Institute, Little Rock, Arkansas
  - University of Colorado Health, Aurora, Colorado
  - University of Florida College of Medicine, Gainesville, Florida
  - Indiana Hemophilia and Thrombosis Center, Indianapolis, Indiana
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
- AKH - Medizinische Universität Wien, Vienna, Austria
- France (5):
  - Hopital Cardiologique - CHU Lille, Lille, Nord
  - Hôpital Necker - Enfants Malades, Paris, Paris
  - Groupement Hospitalier Est- Hôpital Louis Pradel, Bron
  - Groupe Hospitalier Pellegrin - Hôpital Pellegrin, Gironde
  - Groupement Hospitalier Sud - Hôpital Bicêtre, Le Kremlin-Bicêtre
- Germany (2):
  - Klinikum der Johann Wolfgang Goethe-Universitaet, Frankfurt
  - Werlhof-Institut GmbH, Hanover
- Italy (6):
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera Pediatrica Santobono Pausillipon, Napoli
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Azienda Ospedaliera Universitaria Policlinico Umberto I - Università di Roma La Sapienza, Roma
  - Ospedale Pediatrico Bambino Gesù, Roma
- Erasmus Medisch Centrum, Rotterdam, Netherlands
- Russia (2):
  - SAIH "Kemerovo Regional Clinical Hospital", Kemerovo
  - FSBI of Science "Kirov Scientific and Research Institute of Hematology and Blood Transfusion of FMBA, Kirov
- Spain (3):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia
- Turkey (Türkiye) (3):
  - Istanbul University Oncology Institute, Istanbul
  - Ege University Medical Faculty, Izmir
  - Ondokuz Mayis Univ. Med. Fac., Samsun

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fe84db2bf003ab47b19

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 23 investigative sites globally from 1 April 2019 to 30 January 2025.
Pre-assignment Details: A total of 38 participants with diagnosis of Von Willebrand disease were enrolled. Only participants who received treatment in study(N=35) were included in analysis. These participants received recombinant von Willebrand factor (rVWF) [vonicog alfa], 50±10 international units per kilogram (IU/kg),intravenous(IV) infusion in either prophylaxis or on demand cohorts. Some participants received supportive treatment with ADVATE for treating bleeding episodes (BEs) if deemed necessary by investigator.
Groups:
- Cohort 1: Prophylaxis: Adult participants who transitioned from the phase 3 prophylaxis parent study 071301 (NCT02973087) received the same prophylactic dose, 50±10 IU/kg, IV infusion of vonicog alfa twice weekly as in parent study 071301.
- Cohort 2: Prophylaxis: Adult participants who transitioned from parent study 071301 (NCT02973087) with no clinically significant BE for the past 6 months started this continuation study at a lower dose/frequency of vonicog alfa once weekly or twice weekly prophylactic dose, 50±10 IU/kg, IV infusion compared to the dose received (50±10 IU/kg, IV infusion, thrice weekly) in parent study 071301.
- Cohort 3: Prophylaxis: Adolescent participants (aged 12 to less than [<]18 years) who transitioned from the phase 3 OD and surgery parent study 071102 (NCT02932618) switched from receiving vonicog alfa OD treatment to receiving prophylactic dose of vonicog alfa 50±10 IU/kg, IV infusion, once weekly or twice weekly in this continuation study.
- Cohort 4: Prophylaxis: Newly enrolled adult and adolescent (aged 12 to <18 years) participants who switched from OD treatment with Von Willebrand Factor (VWF) products started 50±10 IU/kg, IV infusion once weekly prophylaxis with vonicog alfa in this continuation study.
- Cohort 5: On Demand: Pediatric participants of all ages from parent study 071102 (NCT02932618) continued receiving OD treatment of vonicog alfa 50±10 IU/kg, IV infusion, once weekly or twice weekly in this continuation study.
- Cohort 6: On Demand: Adult participants from parent study 071301 (NCT02973087) switched back from prophylactic treatment in study 071301 to OD treatment of vonicog alfa 50±10 IU/kg, IV infusion, once weekly or twice weekly in this continuation study.
Period: Overall Study
Arm/Group | Cohort 1: Prophylaxis | Cohort 2: Prophylaxis | Cohort 3: Prophylaxis | Cohort 4: Prophylaxis | Cohort 5: On Demand | Cohort 6: On Demand
Started | 10 | 1 | 1 | 5 | 16 | 2
Completed | 10 | 1 | 1 | 3 | 15 | 1
Not Completed | 0 | 0 | 0 | 2 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Site Closed by Sponsor | 0 | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) consisted of all participants who satisfied all entry criteria and received any amount of study drug.
Groups:
- Cohort 3: Prophylaxis: Adolescent participants (aged 12 to <18 years) who transitioned from the phase 3 OD and surgery parent study 071102 (NCT02932618) switched from receiving vonicog alfa OD treatment to receiving prophylactic dose of vonicog alfa 50±10 IU/kg, IV infusion, once weekly or twice weekly in this continuation study.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Prophylaxis | Cohort 2: Prophylaxis | Cohort 3: Prophylaxis | Cohort 4: Prophylaxis | Cohort 5: On Demand | Cohort 6: On Demand | Total
Number analyzed (Participants) | 10 | 1 | 1 | 5 | 16 | 2 | 35
Age, Customized [Count of Participants; unit: Participants] — Population: 2 Participants aged 18 years old in cohort 5 were <18 years of age at the time of enrollment in the parent study 071102 (NCT02932618). They turned 18 years prior to transitioning into this study, their inclusion aligns with the study design, ensuring continuity in cohort assignment, and the age classification at the time of initial enrollment remains relevant for analytical consistency.
  Participants
    <6 years | 0 | 0 | 0 | 0 | 3 | 0 | 3
    >=6 to <12 years | 0 | 0 | 0 | 0 | 5 | 0 | 5
    >=12 to <18 years | 0 | 0 | 1 | 2 | 6 | 0 | 9
    >=18 years | 10 | 1 | 0 | 3 | 2 | 2 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 0 | 2 | 9 | 1 | 17
  Male | 6 | 0 | 1 | 3 | 7 | 1 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1 | 0 | 2
  Not Hispanic or Latino | 8 | 0 | 1 | 5 | 14 | 2 | 30
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 1 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 9 | 0 | 1 | 4 | 14 | 2 | 30
  More than one race | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 0 | 1 | 1 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Spontaneous Annualized Bleeding Rate (sABR)
Description: sABR was derived as [number of treated bleeds] / [duration in years]. Bleeds with unknown causality were considered as spontaneous. Bleeds were categorized based on the investigator assessment of cause. sABR during the first 12 months of prophylactic treatment with rVWF (vonicog alfa) was reported.
Time Frame: Up to 12 months
Population: The FAS consisted of all participants who satisfied all the entry criteria and received any amount of study drug.
Measure: Mean (Standard Deviation); unit: spontaneous bleeds per year
Arm/Group | Cohort 1: Prophylaxis | Cohort 2: Prophylaxis | Cohort 3: Prophylaxis | Cohort 4: Prophylaxis
Number analyzed (Participants) | 10 | 1 | 1 | 5
spontaneous bleeds per year | 1.430 (2.3894) | 1.040 (NA) — Standard deviation was not estimable for a single participant. | 0.000 (NA) — Standard deviation was not estimable for a single participant. | 3.022 (2.4746)

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE): any untoward medical occurrence in a participant administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it is related to medicinal product. TEAE was defined as any AE that started after the first administration of study drug in this continuation study. Serious TEAEs: any untoward medical occurrence that: 1) results in death, 2) is life-threatening, 3) requires inpatient hospitalization or prolongation of existing hospitalization, 4) results in persistent or significant disability/incapacity, 5) leads to a congenital anomaly/birth defect in the offspring of the participant or 6) is medically important.
Time Frame: Up to 5.8 years
Population: The Safety Analysis Set (SAS) consisted of all participants who received any amount of vonicog alfa as obtained from the study drug administration eDiary, study drug administration details eCRF, or PK infusion eCRF.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Prophylaxis | Cohort 2: Prophylaxis | Cohort 3: Prophylaxis | Cohort 4: Prophylaxis | Cohort 5: On Demand | Cohort 6: On Demand
Number analyzed (Participants) | 10 | 1 | 1 | 5 | 16 | 2
Participants
  TEAEs | 8 | 1 | 1 | 4 | 15 | 2
  Serious TEAEs | 3 | 0 | 0 | 1 | 3 | 1

3. Secondary Outcome: Number of Participants Based on Severity of TEAEs
Description: An AE is defined as any untoward medical occurrence in a participant administered IP that does not necessarily have a causal relationship with the treatment. TEAE was defined as any AE that started after the first administration of study drug in this continuation study. Severity of TEAEs was determined by following definitions: Mild: No limitation of usual activities; Moderate: Some limitation of usual activities and may required therapeutic intervention; Severe: Inability to carry out usual activities with sequelae, which required therapeutic intervention. Number of participants with TEAEs based on severity of TEAEs were reported.
Time Frame: Up to 5.8 years
Population: The SAS consisted of all participants who received any amount of vonicog alfa as obtained from the study drug administration eDiary, study drug administration details eCRF, or PK infusion eCRF.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Prophylaxis | Cohort 2: Prophylaxis | Cohort 3: Prophylaxis | Cohort 4: Prophylaxis | Cohort 5: On Demand | Cohort 6: On Demand
Number analyzed (Participants) | 10 | 1 | 1 | 5 | 16 | 2
Participants
  Mild | 7 | 1 | 1 | 4 | 14 | 2
  Moderate | 7 | 0 | 0 | 3 | 11 | 1
  Severe | 3 | 0 | 0 | 1 | 1 | 2

4. Secondary Outcome: Number of Participants Based on Causality of TEAEs
Description: An AE is defined as any untoward medical occurrence in a participant administered IP that does not necessarily have a causal relationship with the treatment. TEAE was defined as any AE that started after the first administration of study drug in this continuation study. A physician/investigator made the assessment of relationship to investigational product for each AE. Number of participants with TEAEs based on causality were reported.
Time Frame: Up to 5.8 years
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Prophylaxis | Cohort 2: Prophylaxis | Cohort 3: Prophylaxis | Cohort 4: Prophylaxis | Cohort 5: On Demand | Cohort 6: On Demand
Number analyzed (Participants) | 10 | 1 | 1 | 5 | 16 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Thromboembolic Events
Description: Thromboembolism defined as formation of a clot (thrombus) in a blood vessel that breaks loose, is carried by the blood stream and could plug another vessel. Number of participants with thromboembolic events as TEAEs of special interest were reported.
Time Frame: Up to 5.8 years
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Prophylaxis | Cohort 2: Prophylaxis | Cohort 3: Prophylaxis | Cohort 4: Prophylaxis | Cohort 5: On Demand | Cohort 6: On Demand
Number analyzed (Participants) | 10 | 1 | 1 | 5 | 16 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Hypersensitivity Reactions
Description: Hypersensitivity (also called hypersensitivity reaction or intolerance) defined as undesirable reactions produced by the normal immune system, including allergies and autoimmunity. Potential hypersensitivity events were identified by broad search criteria and then medically assessed. Number of participants with hypersensitivity reactions as TEAEs of special interest was calculated.
Time Frame: Up to 5.8 years
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Prophylaxis | Cohort 2: Prophylaxis | Cohort 3: Prophylaxis | Cohort 4: Prophylaxis | Cohort 5: On Demand | Cohort 6: On Demand
Number analyzed (Participants) | 10 | 1 | 1 | 5 | 16 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants Who Developed Neutralizing Antibodies to Von Willebrand Factor (VWF)
Description: Three functional VWF assays for von Willebrand factor collagen binding (VWF:CB), von Willebrand factor: Ristocetin Cofactor (VWF:RCo) and von Willebrand factor VIII B (VWF:FVIIIB) were used to test the presence of neutralizing anti-VWF antibodies. Neutralizing antibodies to VWF:RCo, VWF:CB and VWF:FVIIIB activities were measured by assays based on the Bethesda assay established for quantitative analysis of FVIII inhibitors (Nijmegen modification of the Bethesda assay). Only confirmed neutralizing anti -VWF antibodies were considered inhibitors. Number of participants who developed neutralizing antibodies to rVWF were assessed.
Time Frame: Up to 5.8 years
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Prophylaxis | Cohort 2: Prophylaxis | Cohort 3: Prophylaxis | Cohort 4: Prophylaxis | Cohort 5: On Demand | Cohort 6: On Demand
Number analyzed (Participants) | 10 | 1 | 1 | 5 | 16 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants Who Developed Neutralizing Antibodies to Factor VIII (FVIII)
Description: Three functional VWF assays for von Willebrand factor collagen binding (VWF:CB), von Willebrand factor: Ristocetin Cofactor (VWF:RCo) and von Willebrand factor VIII B (VWF:FVIIIB) were used to test the presence of neutralizing anti-VWF antibodies. Neutralizing antibodies to VWF:RCo, VWF:CB and VWF:FVIIIB activities was measured by assays based on the Bethesda assay established for quantitative analysis of FVIII inhibitors (Nijmegen modification of the Bethesda assay). Only confirmed neutralizing anti -VWF antibodies were considered inhibitors. Number of participants who developed neutralizing antibodies to FVIII were assessed.
Time Frame: Up to 5.8 years
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Prophylaxis | Cohort 2: Prophylaxis | Cohort 3: Prophylaxis | Cohort 4: Prophylaxis | Cohort 5: On Demand | Cohort 6: On Demand
Number analyzed (Participants) | 10 | 1 | 1 | 5 | 16 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants Who Developed Total Binding Antibodies to Von Willebrand Factor (VWF)
Description: The presence of total binding anti-VWF antibodies was determined by an enzyme-linked immunosorbent assay (ELISA) employing polyclonal anti-human Immunoglobulin (Ig) antibodies (IgG, IgM and IgA). Number of participants who developed of total binding antibodies to rVWF were assessed.
Time Frame: Up to 5.8 years
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Prophylaxis | Cohort 2: Prophylaxis | Cohort 3: Prophylaxis | Cohort 4: Prophylaxis | Cohort 5: On Demand | Cohort 6: On Demand
Number analyzed (Participants) | 10 | 1 | 1 | 5 | 16 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants Who Developed Total Binding Antibodies to Factor VIII (FVIII)
Description: Binding antibodies against FVIII were analyzed using a proprietary enzyme immunoassay. Number of participants who developed of total binding antibodies to FVIII were assessed.
Time Frame: Up to 5.8 years
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Prophylaxis | Cohort 2: Prophylaxis | Cohort 3: Prophylaxis | Cohort 4: Prophylaxis | Cohort 5: On Demand | Cohort 6: On Demand
Number analyzed (Participants) | 10 | 1 | 1 | 5 | 16 | 2
Participants | 0 | 0 | 0 | 0 | 1 | 0

11. Secondary Outcome: Number of Participants Who Developed Binding Antibodies to Chinese Hamster Ovary (CHO) Proteins
Description: Total Ig antibodies (IgG, IgA, IgM) against CHO protein were analyzed using ELISA. Number of participants who developed binding antibodies to CHO proteins were assessed.
Time Frame: Up to 5.8 years
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Prophylaxis | Cohort 2: Prophylaxis | Cohort 3: Prophylaxis | Cohort 4: Prophylaxis | Cohort 5: On Demand | Cohort 6: On Demand
Number analyzed (Participants) | 10 | 1 | 1 | 5 | 16 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Participants Who Developed Binding Antibodies to Mouse Immunoglobulin G (IgG)
Description: Detection and quantification of IgG antibodies originating from human plasma that were directed against mouse-IgG (HAMA: human anti- mouse antibodies) were assessed using ELISA (Medac, Hamburg, Germany). Number of participants who developed binding antibodies to Mouse IgG were assessed.
Time Frame: Up to 5.8 years
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Prophylaxis | Cohort 2: Prophylaxis | Cohort 3: Prophylaxis | Cohort 4: Prophylaxis | Cohort 5: On Demand | Cohort 6: On Demand
Number analyzed (Participants) | 10 | 1 | 1 | 5 | 16 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Number of Participants Who Develop Binding Antibodies to Recombinant Furin (rFurin)
Description: Total Ig antibodies (IgG, IgA, IgM) against human furin were analyzed using ELISA. Number of participants who developed binding antibodies to rFurin were assessed.
Time Frame: Up to 5.8 years
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Prophylaxis | Cohort 2: Prophylaxis | Cohort 3: Prophylaxis | Cohort 4: Prophylaxis | Cohort 5: On Demand | Cohort 6: On Demand
Number analyzed (Participants) | 10 | 1 | 1 | 5 | 16 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs
Description: Vital signs included blood pressure (systolic and diastolic), pulse rate, respiratory rate and body temperature. Number of participants with clinically significant change from baseline in vital signs were assessed.
Time Frame: Up to 5.8 years
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Prophylaxis | Cohort 2: Prophylaxis | Cohort 3: Prophylaxis | Cohort 4: Prophylaxis | Cohort 5: On Demand | Cohort 6: On Demand
Number analyzed (Participants) | 10 | 1 | 1 | 5 | 16 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Number of Participants With Clinically Significant Changes in Laboratory Parameters
Description: Clinical laboratory parameters included serum chemistry, hematology and urinalysis assessments. Number of participants with clinically significant change from baseline in clinical laboratory parameters were assessed.
Time Frame: Up to 5.8 years
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Prophylaxis | Cohort 2: Prophylaxis | Cohort 3: Prophylaxis | Cohort 4: Prophylaxis | Cohort 5: On Demand | Cohort 6: On Demand
Number analyzed (Participants) | 10 | 1 | 1 | 5 | 16 | 2
Participants
  Serum Chemistry | 0 | 0 | 0 | 0 | 0 | 0
  Hematology | 0 | 0 | 0 | 0 | 0 | 0
  Urinalysis | 0 | 0 | 0 | 0 | NA — No postbaseline results were collected for any urinalysis parameters in the OD cohorts. | NA — No postbaseline results were collected for any urinalysis parameters in the OD cohorts.

16. Secondary Outcome: Spontaneous Annualized Bleeding Rate (sABR) Under Prophylactic Treatment
Description: sABR was derived as [number of treated bleeds] / [duration in years]. Bleeds with unknown causality were considered as spontaneous. Bleeds were categorized based on the investigator assessment of cause. sABR during prophylaxis treatment with rVWF (vonicog alfa) while enrolled in the study were reported.
Time Frame: Up to 5.8 years
Population: The FAS consisted of all participants who satisfied all the entry criteria and received any amount of study drug.
Measure: Mean (Standard Deviation); unit: spontaneous bleeds per year
Arm/Group | Cohort 1: Prophylaxis | Cohort 2: Prophylaxis | Cohort 3: Prophylaxis | Cohort 4: Prophylaxis
Number analyzed (Participants) | 10 | 1 | 1 | 5
spontaneous bleeds per year | 1.122 (2.1084) | 0.330 (NA) — Standard deviation was not estimable for a single participant. | 0.000 (NA) — Standard deviation was not estimable for a single participant. | 2.110 (1.9954)

17. Secondary Outcome: Number of Participants Categorized Based on Weekly Number of Infusions
Description: Categorized as ≥ 0 to < 1 infusion per week, ≥ 1 to < 2 infusions per week, ≥ 2 to < 3 infusions per week, ≥ 3 infusions per week. The number of participants categorized based on number of infusions per week during prophylactic treatment with rVWF (vonicog alfa) were reported.
Time Frame: Up to 5.8 years
Population: The FAS consisted of all participants who satisfied all the entry criteria and received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Prophylaxis | Cohort 2: Prophylaxis | Cohort 3: Prophylaxis | Cohort 4: Prophylaxis
Number analyzed (Participants) | 10 | 1 | 1 | 5
Participants
  ≥0 to <1 | 1 [lower limit 0] | 0 | 0 | 0
  ≥ 1to <2 | 6 [lower limit 60.0] | 1 | 1 | 5
  ≥2 to <3 | 3 [lower limit 40.0] | 0 | 0 | 0
  ≥3 | 0 [lower limit 0] | 0 | 0 | 0

18. Secondary Outcome: Number of Participants Categorized Based on Spontaneous Annualized Bleeding Rate (sABR)
Description: The sABR was the number of spontaneous bleeds divided by the observation period in years, where an observation period = (date of completion/termination-date of first dose+1)/365.2425. sABR was categorized based on number of BEs as 0, greater than (>) 0 through 2, >2 through 5, >5 during the prophylactic treatment with rVWF (vonicog alfa). Bleeding at multiple locations related to the same injury was counted as single BE. BEs of unknown cause were counted as spontaneous bleeds. Number of participants categorized based on sABR during prophylactic treatment with rVWF (vonicog alfa) were reported.
Time Frame: Up to 5.8 years
Population: The FAS consisted of all participants who satisfied all entry criteria and received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Prophylaxis | Cohort 2: Prophylaxis | Cohort 3: Prophylaxis | Cohort 4: Prophylaxis
Number analyzed (Participants) | 10 | 1 | 1 | 5
Participants
  0 bleeds/year | 5 | 0 | 1 | 0
  >0 to ≤2 bleeds/year | 3 | 1 | 0 | 3
  >2 to ≤5 bleeds/year | 1 | 0 | 0 | 1
  >5 bleeds/year | 1 | 0 | 0 | 1

19. Secondary Outcome: Time to First Bleeding Event on Prophylaxis Treatment
Description: Time to event estimates and confidence intervals obtained from Kaplan-Meier analysis. Participants with 0 bleeds during each study period were censored at the date of the last day in that study period.
Time Frame: Up to 5.8 years
Population: The FAS consisted of all participants who satisfied all entry criteria and received any amount of study drug.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Cohort 1: Prophylaxis | Cohort 2: Prophylaxis | Cohort 3: Prophylaxis | Cohort 4: Prophylaxis
Number analyzed (Participants) | 10 | 1 | 1 | 5
days | 172 [5 to NA] — The upper limit of 95% Confidence interval was not estimable due to censoring. | 141 [NA to NA] — The lower and upper limit of 95% Confidence interval was not estimable for a single participant. | NA [NA to NA] — Median was not estimable due to censoring, and the lower and upper limit of 95% Confidence interval was not estimable for a single participant. | 88 [9 to NA] — The upper limit of 95% Confidence interval was not estimable due to censoring.

20. Secondary Outcome: Spontaneous Annualized Bleeding Rate (sABR) by Location of Bleeding
Description: sABR was derived as [number of treated bleeds] / [duration in years]. sABR for BEs based on location of bleeding: Skin, Muscle, Mucosal Nasal, Mucosal Oral, Joint, Gastrointestinal (GI), Menstrual/Heavy Menstrual, Venipuncture Site, Soft Tissue, Body Cavity, Hematuria, Central Nervous System (CNS) and Other, while on prophylactic treatment with rVWF (vonicog alfa) were reported.
Time Frame: Up to 5.8 years
Population: The FAS consisted of all participants who satisfied all entry criteria and received any amount of study drug. Number analyzed is the number of participants with data available for analyses for the specified category.
Measure: Mean (Standard Deviation); unit: bleeds per year
Arm/Group | Cohort 1: Prophylaxis | Cohort 2: Prophylaxis | Cohort 3: Prophylaxis | Cohort 4: Prophylaxis
Number analyzed (Participants) | 10 | 1 | 1 | 5
bleeds per year
  Skin | 0.033 (0.1044) | 0.000 (NA) — Standard deviation was not estimable for a single participant. | 0.000 (NA) — Standard deviation was not estimable for a single participant. | 0.000 (0.0000)
  Muscle | 0.000 (0.0000) | 0.000 (NA) — Standard deviation was not estimable for a single participant. | 0.000 (NA) — Standard deviation was not estimable for a single participant. | 0.068 (0.1521)
  Mucosal, Nasal | 0.199 (0.3542) | 0.000 (NA) — Standard deviation was not estimable for a single participant. | 0.000 (NA) — Standard deviation was not estimable for a single participant. | 0.068 (0.1521)
  Mucosal, Oral | 0.268 (0.7358) | 0.330 (NA) — Standard deviation was not estimable for a single participant. | 0.000 (NA) — Standard deviation was not estimable for a single participant. | 0.268 (0.5993)
  Joint | 0.067 (0.2119) | 0.000 (NA) — Standard deviation was not estimable for a single participant. | 0.000 (NA) — Standard deviation was not estimable for a single participant. | 1.370 (2.3644)
  GI | 0.000 (0.0000) | 0.000 (NA) — Standard deviation was not estimable for a single participant. | 0.000 (NA) — Standard deviation was not estimable for a single participant. | 0.136 (0.3041)
  Menstrual/Heavy Menstrual: number analyzed (Participants) | 2 | 1 | 0 | 2
  Menstrual/Heavy Menstrual | 2.770 (3.9174) | 0.000 (NA) — Standard deviation was not estimable for a single participant. |  | 0.500 (0.7071)
  Venipuncture Site | 0.000 (0.0000) | 0.000 (NA) — Standard deviation was not estimable for a single participant. | 0.000 (NA) — Standard deviation was not estimable for a single participant. | 0.000 (0.0000)
  Soft Tissue | 0.000 (0.0000) | 0.000 (NA) — Standard deviation was not estimable for a single participant. | 0.000 (NA) — Standard deviation was not estimable for a single participant. | 0.000 (0.0000)
  Body Cavity | 0.000 (0.0000) | 0.000 (NA) — Standard deviation was not estimable for a single participant. | 0.000 (NA) — Standard deviation was not estimable for a single participant. | 0.000 (0.0000)
  Hematuria | 0.000 (0.0000) | 0.000 (NA) — Standard deviation was not estimable for a single participant. | 0.000 (NA) — Standard deviation was not estimable for a single participant. | 0.000 (0.0000)
  CNS | 0.000 (0.0000) | 0.000 (NA) — Standard deviation was not estimable for a single participant. | 0.000 (NA) — Standard deviation was not estimable for a single participant. | 0.000 (0.0000)
  Other | 0.067 (0.1413) | 0.000 (NA) — Standard deviation was not estimable for a single participant. | 0.000 (NA) — Standard deviation was not estimable for a single participant. | 0.068 (0.1521)

21. Secondary Outcome: Total Number of Infusions During Prophylactic Treatment
Description: Total number of infusions during prophylactic treatment with rVWF (vonicog alfa) were reported.
Time Frame: Up to 5.8 years
Population: The FAS consisted of all participants who satisfied all the entry criteria and received any amount of study drug.
Measure: Mean (Standard Deviation); unit: infusions
Arm/Group | Cohort 1: Prophylaxis | Cohort 2: Prophylaxis | Cohort 3: Prophylaxis | Cohort 4: Prophylaxis
Number analyzed (Participants) | 10 | 1 | 1 | 5
infusions | 287.8 (53.42) | 157.0 (NA) — Standard deviation was not estimable for a single participant. | 177.0 (NA) — Standard deviation was not estimable for a single participant. | 159.2 (41.55)

22. Secondary Outcome: Average Number of Infusions Per Week During Prophylactic Treatment
Description: Average number of infusions per week during prophylactic treatment with rVWF (vonicog alfa) were reported.
Time Frame: Up to 5.8 years
Population: The FAS consisted of all participants who satisfied all the entry criteria and received any amount of study drug.
Measure: Mean (Standard Deviation); unit: infusions per week
Arm/Group | Cohort 1: Prophylaxis | Cohort 2: Prophylaxis | Cohort 3: Prophylaxis | Cohort 4: Prophylaxis
Number analyzed (Participants) | 10 | 1 | 1 | 5
infusions per week | 1.87 (0.351) | 1.01 (NA) — Standard deviation was not estimable for a single participant. | 1.14 (NA) — Standard deviation was not estimable for a single participant. | 1.38 (0.372)

23. Secondary Outcome: Total Weight Adjusted Consumption of Recombinant Von Willebrand Factor (rVWF) (Vonicog Alfa) Per Participant During Prophylactic Treatment
Description: For each participant, the body weight-adjusted dose (IU/kg) was derived as the number of units of rVWF infused (IU) divided by the last available body weight (kilogram [kg]) prior to the infusion. Total weight adjusted consumption of rVWF (vonicog alfa) per participant during prophylactic treatment with rVWF (vonicog alfa) was reported as International Units per kilogram (IU/kg).
Time Frame: Up to 5.8 years
Population: The FAS consisted of all participants who satisfied all the entry criteria and received any amount of study drug.
Measure: Mean (Standard Deviation); unit: IU/kg
Arm/Group | Cohort 1: Prophylaxis | Cohort 2: Prophylaxis | Cohort 3: Prophylaxis | Cohort 4: Prophylaxis
Number analyzed (Participants) | 10 | 1 | 1 | 5
IU/kg | 14953.497 (3349.4461) | 9992.460 (NA) — Standard deviation was not estimable for a single participant. | 9270.620 (NA) — Standard deviation was not estimable for a single participant. | 9171.746 (1505.5667)

24. Secondary Outcome: Number of Participants Who Achieved Transfusion-free Maintenance of Hemoglobin Levels
Description: Transfusion free maintenance of hemoglobin levels during prophylactic treatment with rVWF (vonicog alfa) were reported.
Time Frame: Up to 5.8 years
Population: The FAS consisted of all participants who satisfied all the entry criteria and received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Prophylaxis | Cohort 2: Prophylaxis | Cohort 3: Prophylaxis | Cohort 4: Prophylaxis
Number analyzed (Participants) | 10 | 1 | 1 | 5
Participants | 8 | 1 | 1 | 5

25. Secondary Outcome: Change From Baseline in Ferritin Levels Over Time
Description: Change from baseline in ferritin levels over time during prophylactic treatment with rVWF (vonicog alfa) were reported. Baseline Ferritin lab assay for rollover participants in cohorts 1, 2 and 3 were not mandatory per protocol at the Screening Visit of this study as the results from End of Study (EOS) visit of parent studies were expected to be utilized for rollover cohorts 1-3. However, many participants in cohort 1 did not have this data collected at EOS Visit of parent study 071301 and no participant in cohorts 2 and 3 had this data collected at EOS Visit of parent studies 071301 and 071102.
Time Frame: Up to 5.8 years
Population: The FAS consisted of all participants who satisfied all the entry criteria and received any amount of study drug. Overall number of participants analyzed is the number of participants with data available for analyses at Baseline. Number analyzed is the number of participants with data available for analyses at the specified timepoint.
Measure: Mean (Standard Deviation); unit: picomole per liter (pmol/L)
Arm/Group | Cohort 1: Prophylaxis | Cohort 2: Prophylaxis | Cohort 3: Prophylaxis | Cohort 4: Prophylaxis
Number analyzed (Participants) | 2 | 0 | 0 | 5
picomole per liter (pmol/L)
  Baseline | 148.5 (171.83) |  |  | 90.8 (110.82)
  Month 1 | 11.0 (18.38) |  |  | -31.0 (44.89)
  Month 2 | 0.0 (1.41) |  |  | -43.8 (59.60)
  Month 3: number analyzed (Participants) | 2 | 0 | 0 | 4
  Month 3 | -18.5 (21.92) |  |  | -33.3 (64.57)
  Month 6 | 2.0 (2.83) |  |  | -16.6 (19.88)
  Month 9 | 58.5 (91.22) |  |  | -12.8 (53.05)
  Month 12: number analyzed (Participants) | 2 | 0 | 0 | 4
  Month 12 | 19.0 (26.87) |  |  | -27.0 (27.51)
  Month 15: number analyzed (Participants) | 2 | 0 | 0 | 3
  Month 15 | 5.5 (13.44) |  |  | -25.7 (80.16)
  Month 18: number analyzed (Participants) | 2 | 0 | 0 | 3
  Month 18 | 18.0 (46.67) |  |  | -49.7 (52.56)
  Month 21 | 37.5 (64.35) |  |  | -59.3 (50.16)
  Month 24 | 12.0 (26.87) |  |  | -53.3 (91.22)
  Month 27 | 34.0 (60.81) |  |  | -54.0 (55.56)
  Month 30: number analyzed (Participants) | 2 | 0 | 0 | 3
  Month 30 | 46.5 (77.07) |  |  | -70.7 (70.12)
  Month 33: number analyzed (Participants) | 2 | 0 | 0 | 3
  Month 33 | 71.5 (106.77) |  |  | -21.3 (114.00)
  End of Study | 38.5 (48.79) |  |  | -27.6 (52.46)

26. Secondary Outcome: Overall Hemostatic Efficacy Rating
Description: Overall Hemostatic Efficacy Rating at resolution of bleed with respect to treatment of BEs for initial 12 months of study in OD cohorts. Hemostatic efficacy for treatment of BEs was rated on 4-point Likert scale as:excellent=full relief of pain&cessation of objective signs of bleeding after single infusion,no additional infusion is required for control of bleeding&administration of further infusion to maintain hemostasis would not affect scoring;good=definite pain relief&/or improvement in signs of bleeding after single infusion,possibly requires >2 infusions for complete resolution&administration of further infusion to maintain hemostasis would not affect scoring;fair=probable&/or slight relief of pain&slight improvement in signs of bleeding after single infusion,required multiple infusions for complete resolution;none=no improvement of signs/symptoms or conditions worsen.Missing=number of unique BEs without any overall hemostatic efficacy rating at resolution of breakthrough BE.
Time Frame: Initial 12 months of study
Population: The FAS consisted of all participants who satisfied all the entry criteria and received any amount of study drug. Overall number of participants analyzed is the number of participants with treated bleeding episodes and overall number of units analyzed is the number of bleeding episodes treated in the initial 12 months of the study.
Measure: Number; unit: bleeding episodes
Units Other Than Participants: bleeding episodes
Arm/Group | Cohort 5: On Demand | Cohort 6: On Demand
Number analyzed (Participants) | 15 | 2
Number analyzed (bleeding episodes) | 76 | 24
bleeding episodes
  Excellent | 74 | 21
  Good | 1 | 0
  Fair | 0 | 0
  None | 0 | 0
  Missing | 1 | 3

27. Secondary Outcome: Number of Infusions of Vonicog Alfa
Description: Number of infusions of rVWF (vonicog alfa) utilized to treat BEs during OD treatment while enrolled in the study were reported.
Time Frame: Up to 5.8 years
Population: The FAS consisted of all participants who satisfied all the entry criteria and received any amount of study drug. Overall number of units analyzed is the number of bleeding episodes treated with vonicog alfa.
Measure: Mean (Standard Deviation); unit: infusions
Units Other Than Participants: bleeding episodes
Arm/Group | Cohort 5: On Demand | Cohort 6: On Demand
Number analyzed (Participants) | 16 | 2
Number analyzed (bleeding episodes) | 167 | 35
infusions | 1.1 (0.65) | 1.2 (0.45)

28. Secondary Outcome: Number of Infusions of ADVATE
Description: Number of infusions of ADVATE (rFVIII, octocog alfa) utilized to treat BEs during OD treatment while enrolled in the study were reported.
Time Frame: Up to 5.8 years
Population: The FAS consisted of all participants who satisfied all the entry criteria and received any amount of study drug. Overall number of participants analyzed is the number of participants with ADVATE-treated bleeding episodes. Overall number of units analyzed is the number of bleeding episodes treated with ADVATE.
Measure: Mean (Standard Deviation); unit: infusions
Units Other Than Participants: bleeding episodes
Arm/Group | Cohort 5: On Demand | Cohort 6: On Demand
Number analyzed (Participants) | 7 | 1
Number analyzed (bleeding episodes) | 46 | 2
infusions | 1.1 (0.25) | 1.0 (0.00)

29. Secondary Outcome: Weight-adjusted Consumption of Vonicog Alfa Per Bleeding Episode
Description: Weight-adjusted consumption (IU/kg) was derived as the total units infused (IU) divided by the last available body weight (kg) prior to the infusion. Weight-adjusted consumption of rVWF (vonicog alfa) per bleeding episode during OD treatment while enrolled in the study were reported.
Time Frame: Up to 5.8 years
Population: The FAS consisted of all participants who satisfied all the entry criteria and received any amount of study drug. Overall number of units analyzed is the number of bleeding episodes treated with vonicog alfa and had consumption data available for analysis of this outcome measure.
Measure: Mean (Standard Deviation); unit: IU/kg per bleeding episode
Units Other Than Participants: bleeding episodes
Arm/Group | Cohort 5: On Demand | Cohort 6: On Demand
Number analyzed (Participants) | 16 | 2
Number analyzed (bleeding episodes) | 165 | 35
IU/kg per bleeding episode | 56.109 (33.1312) | 61.713 (26.6936)

30. Secondary Outcome: Weight-adjusted Consumption of ADVATE Per Bleeding Episode
Description: Weight-adjusted consumption (IU/kg) was derived as the total units infused (IU) divided by the last available body weight (kg) prior to the infusion. Weight-adjusted consumption of ADVATE (rFVIII, octocog alfa) per bleeding episode during OD treatment while enrolled in the study were reported.
Time Frame: Up to 5.8 years
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: IU/kg per bleeding episode
Units Other Than Participants: bleeding episodes
Arm/Group | Cohort 5: On Demand | Cohort 6: On Demand
Number analyzed (Participants) | 7 | 1
Number analyzed (bleeding episodes) | 46 | 2
IU/kg per bleeding episode | 39.217 (11.0752) | 35.175 (2.2274)

ADVERSE EVENTS:
Time Frame: Up to 5.8 years
Description: The SAS consisted of all participants who received any amount of rVWF as obtained from the IP administration eDiary, Study Drug Administration Details eCRF or Pharmacokinetic Infusion eCRF.
Groups:
- Cohort 1: Prophylaxis: Adult ≥18 Years: Adult participants who transitioned from the phase 3 prophylaxis parent study 071301 (NCT02973087) received the same prophylactic dose, 50±10 IU/kg, IV infusion of vonicog alfa twice weekly as in parent study 071301.
- Cohort 2: Prophylaxis: Adult ≥18 Years: Adult participants who transitioned from parent study 071301 (NCT02973087) with no clinically significant BE for the past 6 months started this continuation study at a lower dose/frequency of vonicog alfa once weekly or twice weekly prophylactic dose, 50±10 IU/kg, IV infusion compared to the dose received (50±10 IU/kg, IV infusion, thrice weekly) in parent study 071301.
- Cohort 3: Prophylaxis: Pediatric 12 to <18 Years: Adolescent participants (aged 12 to <18 years) who transitioned from the phase 3 OD and surgery parent study 071102 (NCT02932618) switched from receiving vonicog alfa OD treatment to receiving prophylactic dose of vonicog alfa 50±10 IU/kg, IV infusion, once weekly or twice weekly in this continuation study.
- Cohort 4: Prophylaxis: Pediatric 12 to <18 Years: Newly enrolled adolescent (aged 12 to <18 years) participants who switched from OD treatment with VWF products started 50±10 IU/kg, IV infusion once weekly prophylaxis with vonicog alfa in this continuation study.
- Cohort 4: Prophylaxis: Adult ≥18 Years: Newly enrolled adult participants who switched from OD treatment with VWF products started 50±10 IU/kg, IV infusion once weekly prophylaxis with vonicog alfa in this continuation study.
- Cohort 5: On Demand: Pediatric <6 Years: Pediatric participants of <6 years of age from Parent Study 071102/NCT02932618 continued receiving OD treatment of vonicog alfa 50±10 IU/kg, IV infusion, once weekly or twice weekly in this continuation study.
- Cohort 5: On Demand: Pediatric 6 to <12 Years: Pediatric participants of 6 to <12 years age from parent study 071102 (NCT02932618) continued receiving OD treatment of vonicog alfa 50±10 IU/kg, IV infusion, once weekly or twice weekly in this continuation study.
- Cohort 5: On Demand: Pediatric 12 to <18 Years: Pediatric participants of 12 to <18 years of age from parent study 071102 (NCT02932618) continued receiving OD treatment of vonicog alfa 50±10 IU/kg, IV infusion, once weekly or twice weekly in this continuation study.
- Cohort 5: On Demand: Adult ≥18 Years: Adult Participants from Parent Study 071102/NCT02932618 continued receiving OD treatment of vonicog alfa 50±10 IU/kg, IV infusion, once weekly or twice weekly in this continuation study.
- Cohort 6: On Demand: Adult ≥18 Years: Adult participants from parent study 071301 (NCT02973087) switched back from prophylactic treatment in Study 071301 to OD treatment of vonicog alfa 50±10 IU/kg, IV infusion, once weekly or twice weekly in this continuation study.
Arm/Group | Cohort 1: Prophylaxis: Adult ≥18 Years | Cohort 2: Prophylaxis: Adult ≥18 Years | Cohort 3: Prophylaxis: Pediatric 12 to <18 Years | Cohort 4: Prophylaxis: Pediatric 12 to <18 Years | Cohort 4: Prophylaxis: Adult ≥18 Years | Cohort 5: On Demand: Pediatric <6 Years | Cohort 5: On Demand: Pediatric 6 to <12 Years | Cohort 5: On Demand: Pediatric 12 to <18 Years | Cohort 5: On Demand: Adult ≥18 Years | Cohort 6: On Demand: Adult ≥18 Years
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/1 | 0/1 | 0/2 | 0/3 | 0/3 | 0/5 | 0/6 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 3/10 | 0/1 | 0/1 | 0/2 | 1/3 | 2/3 | 1/5 | 0/6 | 0/2 | 1/2
Other Adverse Events (participants affected / at risk) | 8/10 | 1/1 | 1/1 | 2/2 | 2/3 | 3/3 | 5/5 | 6/6 | 1/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Prophylaxis: Adult ≥18 Years (N=10) | Cohort 2: Prophylaxis: Adult ≥18 Years (N=1) | Cohort 3: Prophylaxis: Pediatric 12 to <18 Years (N=1) | Cohort 4: Prophylaxis: Pediatric 12 to <18 Years (N=2) | Cohort 4: Prophylaxis: Adult ≥18 Years (N=3) | Cohort 5: On Demand: Pediatric <6 Years (N=3) | Cohort 5: On Demand: Pediatric 6 to <12 Years (N=5) | Cohort 5: On Demand: Pediatric 12 to <18 Years (N=6) | Cohort 5: On Demand: Adult ≥18 Years (N=2) | Cohort 6: On Demand: Adult ≥18 Years (N=2)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronavirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Medical device site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Prophylaxis: Adult ≥18 Years (N=10) | Cohort 2: Prophylaxis: Adult ≥18 Years (N=1) | Cohort 3: Prophylaxis: Pediatric 12 to <18 Years (N=1) | Cohort 4: Prophylaxis: Pediatric 12 to <18 Years (N=2) | Cohort 4: Prophylaxis: Adult ≥18 Years (N=3) | Cohort 5: On Demand: Pediatric <6 Years (N=3) | Cohort 5: On Demand: Pediatric 6 to <12 Years (N=5) | Cohort 5: On Demand: Pediatric 12 to <18 Years (N=6) | Cohort 5: On Demand: Adult ≥18 Years (N=2) | Cohort 6: On Demand: Adult ≥18 Years (N=2)
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Angular cheilitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anti factor VIII antibody positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Astigmatism (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bone contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bundle branch block right (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 1 | 0 | 2 | 3 | 1 | 3 | 1 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronavirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 0
Croup infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Device malfunction (Product Issues) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fracture displacement (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemobilia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemophilic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site rash (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Lymphatic malformation (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Serum ferritin decreased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stress fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth deposit (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tracheobronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 1 | 1
Varicose vein (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Viral rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Zinc deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-12-20): https://cdn.clinicaltrials.gov/large-docs/35/NCT03879135/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-03): https://cdn.clinicaltrials.gov/large-docs/35/NCT03879135/SAP_001.pdf